CLINICAL TRIAL: NCT01438320
Title: A Phase 1 Study of Quercetin in Patients With Hepatitis C
Brief Title: Q-Trial in Patients With Hepatitis C
Acronym: Q
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: American Association for Cancer Research (Other); Tower Cancer Research Foundation (Unknown); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, SAMUEL FRENCH, Assistant Professor, University of California, Los Angeles
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IRB#10-04-063-01; 1R01DK090794-01A1 (NIH)
Record Dates: First submitted 2011-09-14; First posted 2011-09-22 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Hepatitis C
Keywords: Treatment naive; Contraindications to standard therapies; Alternative hepatitis C therapy
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Quercetin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Quercetin (Experimental): Quercetin is a bioflavonoid.
  Interventions: Dietary Supplement: Quercetin

INTERVENTIONS:
Dietary Supplement: Quercetin — Bioflavonoid

SUMMARY:
The goal of this study is to translate laboratory findings that Quercetin, a bioflavonoid, is safe and has antiviral activity in people with hepatitis C.

DETAILED DESCRIPTION:
Chronic hepatitis C (HCV) is a serious chronic condition in the United States affecting millions of people and is the cause of rates of hepatocellular carcinoma recently doubling in the US. Treatment of hepatitis C is proven to be an effective secondary prevention of liver cancer. Current standard antiviral treatments exclude 70-80% of hepatitis C patients from therapies due to intolerable side effects. Our laboratory efforts identified a potential novel approach to hepatitis C treatment and hepatocellular carcinoma prevention with Quercetin, a heat shock protein inhibitor.

This is a Phase I study evaluating the safety and tolerability of Quercetin in hepatitis C patients who have contraindications to standard antiviral treatment (both treatment naïve patients who decline standard therapy, patients who previously had standard treatments with relapse, as well as those who had intolerable side effects previously). The investigators recently demonstrated that the flavonoid Quercetin inhibits hepatitis C viral production in tissue culture, at least partially through its inhibition of heat shock protein expression. This represents a novel mechanism for treating hepatitis C infection. Quercetin also has low toxicity. These promising characteristics motivate the proposed Phase I study. Patients will be recruited through the UCLA Pfleger Liver Institute and treated on an outpatient basis. Toxicity will be closely monitored and reported. Viral load response will be evaluated as a secondary endpoint. The anticipated total number of patients enrolled in the trial will be 20. All patients will be followed for 8 months after taking this first dose of study medication. Patients exhibiting a viral load response will have extended follow-up, ranging from a total follow-up of 12-24 months, to determine persistence of this response.

ELIGIBILITY:
Inclusion Criteria:

* All participants will have detectable HCV RNA in serum; stable viral load within the previous year (no fluctuation > 2 log scale).
* All participants are either treatment-naïve and unwilling to be treated with standard HCV therapies, or were not able to tolerate hepatitis C antiviral due to side effects and completed treatment more than 6 months prior to enrollment into our trial.
* Age range will be from 18-65 years old
* ECOG performance status <2 (Karnofsky >60%)
* Life expectancy of greater than 12 months
* Participants must have:

  * leukocytes >3,000/mcL
  * absolute neutrophil count >1,500/mm(3)
  * hemoglobin >13 or >12 g/dL for men/women
  * platelets >125,000 K/mm(3)
  * total bilirubin <1.5 g/dL
  * AST(SGOT)/ALT(SGPT) <10 X institutional upper limit of normal
  * Albumin >3.4g/dL
  * INR <1.2
  * Alpha Feto-protein <50 ng/mL
  * creatinine within normal institutional limits OR
  * creatinine clearance >60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
* All participants must exhibit the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who are currently on interferon +/- ribavirin or any other anti-viral therapies are excluded from our study. Participants who have previously been treated with hepatitis C antiviral therapy must have recovered from any adverse events due to the agent(s) administered. In addition, their last antiviral therapy must be more than six months prior to their enrollment in our study
* Participants may not be receiving any other investigational agents
* Participants with decompensated liver disease or cirrhosis will be excluded from this trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Quercetin or any bioflavonoid agent
* According to a monogram published by the Natural Medicines Comprehensive Database, drug interactions with Quercetin have been reported to occur with quinolone antibiotics and inhibition of p-glycoprotein or various cytochrome P450 enzymes including CYP3A4/ CYP2C8/ CYP2C9/ CYP2D6. Quercetin interactions with drugs can be categorized into (1) moderate interaction to be avoided based on healthy volunteer studies and (2) moderate interaction to be monitored closely based on in vitro studies demonstrating potential theoretical reduced elimination and increased effects. Screening will be performed prior to treatment.
* Participants with concurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, untreated/active cardiac arrhythmia, psychiatric illness, active moderate alcohol use, or any social situation that would limit compliance with study protocol will be excluded from our study.
* In addition, participants with any other known hepatitis etiologies (hepatitis B co-infection, hemochromatosis, alpha-1 antitrypsin deficiency, Wilson Disease, autoimmune hepatitis, alcohol, drug, obesity induced liver disease); or those with hepatocellular carcinoma will be excluded from this study.
* Pregnant women are excluded from this study.
* Human immunodeficiency virus (HIV)-positive subjects are excluded from our study.
* In addition to renal and hepatic laboratory requirements listed above, renal and liver transplant recipients will be excluded from our study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Adverse Event Score Assessment of Quercetin Given over 28 days in hepatitis C patients who have contraindications to standard antiviral treatment | up to 32 weeks
  Primary outcome for the study will be safety. The investigators will track various laboratory parameters including viral loads and see patients every 2 weeks during our drug phase which is 28 days. After that follow patients every month to see how long antiviral activity will persist if we do see a positive outcome.

SECONDARY OUTCOMES:
Hepatitis C Viral Load Assessment with Quercetin Given Over 28 days | 28 days during drug phase. Possibly this could go further for 32 weeks.
  Hepatitis C viral load will be monitored every 2 wks during the first 28 days when patients are taking Quercetin. After this period, if there is a positive antiviral activity that is seen, we continue to monitor viral load every month to see how long this effect will last.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel W French, MD/PhD, Principal Investigator — University of California, Los Angeles; Nu Lu, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Jonsson Comprehensive Cancer Center. Factor Building, Los Angeles, California, United States

REFERENCES:
- [Background] Gonzalez O, Fontanes V, Raychaudhuri S, Loo R, Loo J, Arumugaswami V, Sun R, Dasgupta A, French SW. The heat shock protein inhibitor Quercetin attenuates hepatitis C virus production. Hepatology. 2009 Dec;50(6):1756-64. doi: 10.1002/hep.23232. PMID 19839005
- [Derived] Lu NT, Crespi CM, Liu NM, Vu JQ, Ahmadieh Y, Wu S, Lin S, McClune A, Durazo F, Saab S, Han S, Neiman DC, Beaven S, French SW. A Phase I Dose Escalation Study Demonstrates Quercetin Safety and Explores Potential for Bioflavonoid Antivirals in Patients with Chronic Hepatitis C. Phytother Res. 2016 Jan;30(1):160-8. doi: 10.1002/ptr.5518. Epub 2015 Dec 1. PMID 26621580
- See also: Media Release regarding exciting in-vitro study of Quercetin against hepatitis C — http://www.sciencedaily.com/releases/2011/04/110412201709.htm